CLINICAL TRIAL: NCT01163851
Title: A Phase 1 Study Evaluating The Pharmacokinetics And Pharmacodynamics Of Rn316 In Combination With Atorvastatin In Hypercholesterolemic Subjects
Brief Title: Pharmacokinetic And Pharmacodynamic Study Of A Single-Dose Of PF-04950615 (RN316) In Combination With Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1481003
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: Hypercholesterolemia; Dyslipidemia; LDL; Cholesterol; High Cholesterol; PF-04950615; RN316
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — bococizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04950615 (RN316) (Experimental)
  Interventions: Biological: 4 mg/kg; Biological: 0.5 mg/kg

INTERVENTIONS:
Biological: 4 mg/kg — RN316 10 mg/ml vial sd. Infusion based on weight Infusion duration = 60 minutes.
  Other Names: PF-04950615 (RN316)
Biological: 0.5 mg/kg — RN316 10 mg/ml vial sd. Infusion based on weight Infusion duration = 60 minutes.
  Other Names: PF-04950615 (RN316)

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics and pharmacodynamics of a single dose of PF-04950615 (RN316) in volunteers on stable doses of atorvastatin. PF-04950615 (RN316) is an investigational drug that is currently being studies as a cholesterol lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* On stable doses of atorvastatin (40 mg daily) for 45 days prior to Day 1.
* BMI 18.5 to 40 kg/m2 inclusive, and body weight equal or lower than 150 kg.

Exclusion Criteria:

* History of a cardiovascular event (e.g., MI ) during the past year.
* Poorly controlled Type 1 or Type 2 Diabetes mellitus (definition: uncontrolled diabetes is defined as HBIAc >9%).
* Poorly controlled hypertension (uncontrolled hypertension is defined as a systolic blood pressure greater than 140 mm Hg or a diastolic blood pressure greater than 90 mm Hg, even with treatment). Subjects who have hypertension and are controlled on stable dosages of anti-hypertensive medications can be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Premier Research Group, Limited, Peoria, Arizona
  - Dedicated Phase 1, Inc., Phoenix, Arizona
  - Premier Research Group Limited, Phoenix, Arizona
  - Vince and Associates Clinical Research, Overland Park, Kansas

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Udata C, Garzone PD, Gumbiner B, Joh T, Liang H, Liao KH, Williams JH, Meng X. A Mechanism-Based Pharmacokinetic/Pharmacodynamic Model for Bococizumab, a Humanized Monoclonal Antibody Against Proprotein Convertase Subtilisin/Kexin Type 9, and Its Application in Early Clinical Development. J Clin Pharmacol. 2017 Jul;57(7):855-864. doi: 10.1002/jcph.867. Epub 2017 Feb 9. PMID 28181260
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481003&StudyName=Pharmacokinetic%20And%20Pharmacodynamic%20Study%20Of%20A%20Single-Dose%20Of%20PF-04950615%20%28RN316%29%20In%20Combination%20with%20Atorvastatin

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04950615 (RN316) 4 mg/kg + Atorvastatin: Participants received single intravenous infusion dose of PF-04950615 (RN316) 4 milligram per kilogram (mg/kg) on Day 4 along with sponsor provided atorvastatin 40 milligram (mg) tablet orally once daily from Day 1 to 7. Participants were on self-administered stable atorvastatin therapy, 40 mg orally once daily prior to Day 1 and after treatment phase (Day 7). Participants were followed up to Day 64.
- PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin: Participants received single intravenous infusion dose of PF-04950615 (RN316) 0.5 mg/kg on Day 4 along with sponsor provided atorvastatin 40 mg tablet orally once daily from Day 1 to 7. Participants were on self-administered stable atorvastatin therapy, 40 mg orally once daily prior to Day 1 and after treatment phase (Day 7). Participants were followed up to Day 64.
Period: Overall Study
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Started | 13 | 12
Treated | 12 | 12
Completed | 12 | 11
Not Completed | 1 | 1
Not completed — Site Closure | 0 | 1
Not completed — Enrolled but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who met the study enrollment criteria and received any amount of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-04950615
Time Frame: 0 (pre-dose on Day 4), 1, 4, 8 and 12 hours (hrs) post intravenous PF-04950615 (RN316) dose, pre atorvastatin dose on Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Population: Pharmacokinetic (PK) parameter analysis population included all enrolled participants who were treated and had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter | 17950000 (2779600) | 933800 (376350)

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04950615
Time Frame: as for outcome 1
Population: PK parameter analysis population included all enrolled participants who were treated and had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
hour | 2.59 [1.00 to 12.10] | 4.00 [1.00 to 7.92]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04950615
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
nanogram per milliliter | 105000 (16587) | 14030 (1680)

4. Primary Outcome: Plasma Decay Half-Life (t1/2) of PF-04950615
Description: Plasma decay half-life is the time measured for the plasma concentration of PF-04950615 to decrease by one half.
Time Frame: as for outcome 1
Population: PK parameter analysis population included all enrolled participants who were treated and had at least 1 of the PK parameters of interest. Here, 'Overall number of participants analyzed' signifies those participants who were evaluable for this measure for each group respectively.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 11 | 7
hour | 157.50 (33.22) | 61.00 (8.89)

5. Primary Outcome: Systemic Clearance (CL) of PF-04950615
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: liter per hour
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 11 | 7
liter per hour | 0.0185 (0.0041) | 0.0392 (0.0031)

6. Primary Outcome: Volume of Distribution at Steady State (Vss) of PF-04950615
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: liter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 11 | 7
liter | 4.248 (1.099) | 3.436 (0.583)

7. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) of PF-04950615
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 11 | 7
nanogram*hour per milliliter | 17960000 (2828500) | 1094000 (123640)

8. Primary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of Atorvastatin
Description: AUCtau was the AUC from time 0 to the end of the dosing interval, where the dosing interval was 12 hours.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 and 12 hrs post-dose on Day 4
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
nanogram*hour per milliliter | 71.73 (32.22) | 89.17 (33.25)

9. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Atorvastatin
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 and 12 hrs post-dose on Day 4, pre atorvastatin dose on Day 5, 6 and 7
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
hour | 1.16 [0.50 to 3.00] | 1.00 [0.50 to 3.02]

10. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Atorvastatin
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 and 12 hrs post-dose on Day 4, pre atorvastatin dose on Day 5, 6 and 7
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
nanogram per milliliter | 15.79 (8.81) | 20.68 (10.58)

11. Primary Outcome: Plasma Decay Half-Life (t1/2) of Atorvastatin
Description: Plasma decay half-life is the time measured for the plasma concentration of atorvastatin to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 and 12 hrs post-dose on Day 4, pre atorvastatin dose on Day 5, 6 and 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 10 | 11
hour | 5.12 (1.38) | 5.09 (0.74)

12. Primary Outcome: Apparent Oral Clearance (CL/F) of Atorvastatin
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 and 12 hrs post-dose on Day 4
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: liter per hour
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
liter per hour | 557.50 (238.33) | 448.70 (196.91)

13. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Atorvastatin
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 and 12 hrs post-dose on Day 4
Population: PK parameter analysis population included all enrolled participants who were treated and had at least 1 of the PK parameters of interest. Here, 'Overall number of participants analyzed' is signifying those participants who were evaluable for this measure for each group respectively.
Measure: Geometric Mean (Standard Deviation); unit: liter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 10 | 11
liter | 3950 (1952.8) | 3353 (1960.8)

14. Secondary Outcome: Change From Baseline in Fasting Low Density Lipoprotein-Cholesterol (LDL-C) at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: Pharmacodynamic analysis population included all enrolled participants who received any amount of study medication and had at least 1 pharmacodynamic parameter of interest. Here, 'Number Participants Analyzed' is signifying those participants who were evaluable for particular category for each arm group respectively.
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
milligram per deciliter
  Change at Day 5 | -14.30 (17.79) | -16.2 (11.56)
  Change at Day 6: number analyzed (Participants) | 11 | 11
  Change at Day 6 | -28.50 (17.22) | -34.00 (19.13)
  Change at Day 7: number analyzed (Participants) | 11 | 11
  Change at Day 7 | -33.30 (22.42) | -47.20 (20.66)
  Change at Day 15: number analyzed (Participants) | 10 | 12
  Change at Day 15 | -52.40 (35.31) | -25.90 (31.94)
  Change at Day 22: number analyzed (Participants) | 9 | 12
  Change at Day 22 | -57.20 (30.71) | 2.10 (36.01)
  Change at Day 29: number analyzed (Participants) | 9 | 12
  Change at Day 29 | -56.90 (35.21) | 9.40 (33.12)
  Change at Day 36 | -55.50 (23.64) | 3.40 (33.09)
  Change at Day 43 | -32.30 (15.64) | 8.80 (34.18)
  Change at Day 50 | -11.40 (13.27) | 4.10 (29.02)
  Change at Day 57: number analyzed (Participants) | 11 | 11
  Change at Day 57 | -1.50 (22.25) | 10.90 (35.79)
  Change at Day 64 | 6.20 (24.62) | 12.10 (33.42)

15. Secondary Outcome: Change From Baseline in Fasting Total Cholesterol at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
milligram per deciliter
  Change at Day 5 | -13.90 (19.48) | -21.60 (15.04)
  Change at Day 6 | -33.30 (19.04) | -38.30 (18.03)
  Change at Day 7 | -37.30 (25.72) | -50.00 (20.50)
  Change at Day 15 | -58.00 (39.02) | -24.30 (38.29)
  Change at Day 22 | -61.30 (34.91) | 7.50 (38.05)
  Change at Day 29 | -62.60 (32.81) | 8.40 (36.28)
  Change at Day 36 | -56.30 (28.61) | 5.30 (36.43)
  Change at Day 43 | -28.90 (19.61) | 9.80 (38.40)
  Change at Day 50 | -6.30 (18.51) | 4.80 (34.39)
  Change at Day 57: number analyzed (Participants) | 12 | 11
  Change at Day 57 | 9.30 (31.92) | 18.50 (34.69)
  Change at Day 64 | 12.10 (23.00) | 15.10 (31.48)

16. Secondary Outcome: Change From Baseline in Fasting Non High-density Lipoprotein-Cholesterol (Non-HDL-C) at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
milligram per deciliter
  Change at Day 5 | 12.60 (21.90) | -19.40 (15.16)
  Change at Day 6 | -31.20 (20.31) | -35.90 (22.27)
  Change at Day 7 | -36.40 (24.50) | -47.60 (24.04)
  Change at Day 15 | -62.50 (39.40) | -30.10 (36.18)
  Change at Day 22 | -68.80 (32.78) | 4.70 (40.14)
  Change at Day 29 | -69.00 (35.01) | 7.90 (39.76)
  Change at Day 36 | -60.00 (29.56) | 3.50 (41.05)
  Change at Day 43 | -35.00 (18.14) | 6.60 (38.85)
  Change at Day 50 | -9.00 (17.87) | 3.10 (37.89)
  Change at Day 57: number analyzed (Participants) | 12 | 11
  Change at Day 57 | 6.50 (32.76) | 14.30 (39.36)
  Change at Day 64 | 12.10 (20.13) | 12.70 (35.12)

17. Secondary Outcome: Change From Baseline in Fasting Triglycerides at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
milligram per deciliter
  Change at Day 5 | 9.20 (61.82) | -15.80 (38.46)
  Change at Day 6 | 11.70 (24.23) | -9.90 (31.22)
  Change at Day 7 | 8.10 (38.09) | -6.90 (44.25)
  Change at Day 15 | -19.60 (41.40) | -21.10 (56.39)
  Change at Day 22 | -4.30 (45.63) | 13.60 (52.71)
  Change at Day 29 | -17.40 (21.51) | -8.20 (60.64)
  Change at Day 36 | -22.20 (54.24) | -0.30 (70.24)
  Change at Day 43 | -13.10 (42.48) | -10.90 (64.52)
  Change at Day 50 | 11.60 (57.86) | -4.90 (79.62)
  Change at Day 57: number analyzed (Participants) | 12 | 11
  Change at Day 57 | 26.20 (63.42) | 16.50 (56.65)
  Change at Day 64 | 29.60 (53.23) | 3.10 (31.78)

18. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein B (ApoB) at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
milligram per deciliter
  Change at Day 5 | -10.90 (7.48) | -13.10 (8.49)
  Change at Day 6 | -22.10 (10.05) | -24.90 (12.88)
  Change at Day 7 | -28.30 (12.57) | -29.50 (16.75)
  Change at Day 15 | -41.90 (19.41) | -21.70 (19.84)
  Change at Day 22 | -44.00 (17.67) | -3.30 (18.78)
  Change at Day 29 | -45.80 (17.61) | -1.10 (23.99)
  Change at Day 36 | -41.10 (15.09) | -2.70 (19.76)
  Change at Day 43 | -27.30 (7.48) | -0.60 (18.47)
  Change at Day 50 | -10.40 (10.53) | -4.60 (20.74)
  Change at Day 57: number analyzed (Participants) | 12 | 11
  Change at Day 57 | -5.10 (15.70) | 4.70 (15.51)
  Change at Day 64 | 2.30 (10.70) | 5.80 (20.99)

19. Secondary Outcome: Change From Baseline in Fasting Apolipoprotein A1 (ApoA1) at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 (RN316) administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
milligram per deciliter
  Change at Day 5 | -3.00 (10.95) | 2.80 (8.70)
  Change at Day 6 | -1.70 (10.79) | -5.60 (8.07)
  Change at Day 7 | 3.40 (10.93) | -1.50 (9.22)
  Change at Day 15 | 6.80 (8.30) | 12.10 (18.48)
  Change at Day 22 | 5.70 (11.13) | 16.10 (18.71)
  Change at Day 29 | 7.50 (13.43) | 11.40 (27.34)
  Change at Day 36 | 10.30 (10.87) | 11.50 (15.09)
  Change at Day 43 | 7.80 (10.73) | 14.90 (15.96)
  Change at Day 50 | 6.50 (8.64) | 5.20 (22.03)
  Change at Day 57: number analyzed (Participants) | 12 | 11
  Change at Day 57 | 4.40 (11.77) | 24.50 (12.51)
  Change at Day 64 | 0.50 (10.82) | 22.10 (19.44)

20. Secondary Outcome: Change From Baseline in Fasting High-Density Lipoprotein (HDL) Cholesterol at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milligram per deciliter
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
milligram per deciliter
  Change at Day 5 | -1.30 (5.60) | -2.20 (7.95)
  Change at Day 6 | -2.10 (4.16) | -2.40 (11.71)
  Change at Day 7 | -0.90 (4.41) | -2.40 (12.63)
  Change at Day 15 | 4.50 (8.01) | 5.90 (5.13)
  Change at Day 22 | 6.70 (4.65) | 2.80 (5.41)
  Change at Day 29 | 6.50 (6.53) | 0.50 (5.99)
  Change at Day 36 | 3.80 (5.52) | 1.90 (8.20)
  Change at Day 43 | 6.10 (6.59) | 3.10 (5.39)
  Change at Day 50 | 2.80 (6.27) | 1.70 (7.71)
  Change at Day 57: number analyzed (Participants) | 12 | 11
  Change at Day 57 | 2.70 (5.26) | 4.20 (9.22)
  Change at Day 64 | -0.0 (6.02) | 2.40 (7.95)

21. Secondary Outcome: Percent Change From Baseline in Fasting Low Density Lipoprotein-Cholesterol (LDL-C) at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
percent change
  Percent change at Day 5 | -15.70 (23.36) | -27.30 (23.60)
  Percent change at Day 6: number analyzed (Participants) | 11 | 11
  Percent change at Day 6 | -33.80 (20.61) | -47.00 (30.57)
  Percent change at Day 7: number analyzed (Participants) | 11 | 11
  Percent change at Day 7 | -38.90 (24.15) | -65.10 (31.82)
  Percent change at Day 15: number analyzed (Participants) | 10 | 12
  Percent change at Day 15 | -61.10 (31.98) | -33.30 (29.80)
  Percent change at Day 22: number analyzed (Participants) | 9 | 12
  Percent change at Day 22 | -71.60 (21.89) | 11.40 (46.23)
  Percent change at Day 29: number analyzed (Participants) | 9 | 12
  Percent change at Day 29 | -68.70 (22.20) | 21.60 (46.26)
  Percent change at Day 36 | -68.20 (15.59) | 14.90 (36.90)
  Percent change at Day 43 | -41.80 (18.87) | 19.70 (38.86)
  Percent change at Day 50 | -14.70 (17.10) | 13.70 (37.36)
  Percent change at Day 57: number analyzed (Participants) | 11 | 11
  Percent change at Day 57 | 1.40 (24.80) | 23.60 (47.93)
  Percent change at Day 64 | 13.40 (31.22) | 25.60 (42.94)

22. Secondary Outcome: Percent Change From Baseline in Total Cholesterol at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
percent change
  Percent change at Day 5 | -8.30 (11.81) | -14.60 (8.87)
  Percent change at Day 6 | -21.20 (10.16) | -26.20 (10.56)
  Percent change at Day 7 | -23.10 (14.16) | -34.10 (11.39)
  Percent change at Day 15 | -35.40 (19.65) | -14.40 (18.89)
  Percent change at Day 22 | -38.40 (16.70) | 7.40 (21.95)
  Percent change at Day 29 | -39.40 (14.50) | 7.40 (19.86)
  Percent change at Day 36 | -36.30 (14.00) | 7.00 (21.50)
  Percent change at Day 43 | -18.90 (10.34) | 9.00 (21.22)
  Percent change at Day 50 | -3.70 (11.17) | 6.00 (19.62)
  Percent change at Day 57: number analyzed (Participants) | 12 | 11
  Percent change at Day 57 | 7.50 (19.31) | 14.30 (20.05)
  Percent change at Day 64 | 10.10 (14.86) | 12.50 (18.07)

23. Secondary Outcome: Percent Change From Baseline in Fasting Non-High-density Lipoprotein-cholesterol (Non-HDL-C) at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
percent change
  Percent change at Day 5 | -9.90 (20.47) | -20.30 (15.38)
  Percent change at Day 6 | -28.70 (16.69) | -37.60 (26.74)
  Percent change at Day 7 | -32.80 (18.81) | -50.00 (26.78)
  Percent change at Day 15 | -56.00 (26.05) | -25.40 (26.16)
  Percent change at Day 22 | -63.90 (18.00) | 14.70 (40.72)
  Percent change at Day 29 | -63.90 (17.86) | 16.10 (40.69)
  Percent change at Day 36 | -57.30 (16.60) | 14.00 (36.59)
  Percent change at Day 43 | -35.70 (16.64) | 14.30 (35.80)
  Percent change at Day 50 | -9.40 (16.55) | 12.90 (38.29)
  Percent change at Day 57: number analyzed (Participants) | 12 | 11
  Percent change at Day 57 | 7.80 (26.93) | 23.80 (44.36)
  Percent change at Day 64 | 15.60 (20.30) | 21.20 (35.27)

24. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides Values at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 (RN316) administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
percent change
  Percent change at Day 5 | 11.20 (65.46) | -3.30 (24.88)
  Percent change at Day 6 | 7.40 (20.29) | 1.10 (22.05)
  Percent change at Day 7 | 5.00 (21.20) | 0.50 (27.67)
  Percent change at Day 15 | -6.10 (41.62) | -1.40 (35.76)
  Percent change at Day 22 | -2.20 (30.73) | 19.90 (42.17)
  Percent change at Day 29 | -14.60 (20.02) | 0.80 (34.11)
  Percent change at Day 36 | -15.90 (32.23) | 12.20 (45.69)
  Percent change at Day 43 | -7.90 (25.94) | 3.20 (33.05)
  Percent change at Day 50 | 12.60 (42.61) | 12.10 (49.12)
  Percent change at Day 57: number analyzed (Participants) | 12 | 11
  Percent change at Day 57 | 20.10 (45.52) | 22.20 (41.65)
  Percent change at Day 64 | 28.60 (42.51) | 7.60 (30.24)

25. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein B (ApoB) Values at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 (RN316) administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
percent change
  Percent change at Day 5 | -13.50 (9.25) | -17.10 (11.22)
  Percent change at Day 6 | -26.90 (11.01) | -31.10 (13.84)
  Percent change at Day 7 | -33.80 (12.27) | -36.10 (15.68)
  Percent change at Day 15 | -48.60 (13.82) | -24.80 (18.18)
  Percent change at Day 22 | -51.50 (11.04) | -0.70 (19.21)
  Percent change at Day 29 | -53.70 (10.37) | 3.80 (26.31)
  Percent change at Day 36 | -48.80 (9.97) | 1.50 (22.64)
  Percent change at Day 43 | -33.80 (8.98) | 2.70 (18.81)
  Percent change at Day 50 | -13.70 (13.70) | -1.50 (21.38)
  Percent change at Day 57: number analyzed (Participants) | 12 | 11
  Percent change at Day 57 | -5.80 (18.03) | 9.40 (19.89)
  Percent change at Day 64 | 3.00 (12.82) | 11.50 (25.50)

26. Secondary Outcome: Percent Change From Baseline in Fasting High-Density Lipoprotein (HDL) Cholesterol Values at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
percent change
  Percent change at Day 5 | -2.50 (11.27) | -1.70 (10.93)
  Percent change at Day 6 | -3.60 (8.24) | -0.90 (18.31)
  Percent change at Day 7 | -1.10 (9.29) | -0.90 (18.01)
  Percent change at Day 15 | 11.10 (19.48) | 13.40 (12.40)
  Percent change at Day 22 | 13.90 (9.65) | 8.00 (11.23)
  Percent change at Day 29 | 14.00 (15.04) | 3.00 (11.72)
  Percent change at Day 36 | 7.80 (11.50) | 7.50 (17.15)
  Percent change at Day 43 | 14.50 (15.67) | 8.70 (8.79)
  Percent change at Day 50 | 6.10 (13.89) | 6.70 (14.20)
  Percent change at Day 57: number analyzed (Participants) | 12 | 11
  Percent change at Day 57 | 6.10 (11.93) | 14.00 (19.37)
  Percent change at Day 64 | 0.50 (12.37) | 8.20 (12.15)

27. Secondary Outcome: Percent Change From Baseline in Fasting Apolipoprotein A1 (ApoA1) Values at Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57 and 64
Description: Baseline value calculated as average of Day 2 and Day 4 measurements prior to PF-04950615 (RN316) administration.
Time Frame: Baseline, Day 5, 6, 7, 15, 22, 29, 36, 43, 50, 57, 64
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
percent change
  Percent change at Day 5 | -1.90 (7.48) | 2.10 (6.61)
  Percent change at Day 6 | -1.00 (7.27) | -4.20 (6.80)
  Percent change at Day 7 | 2.90 (7.14) | -0.80 (7.97)
  Percent change at Day 15 | 5.10 (6.31) | 9.10 (12.52)
  Percent change at Day 22 | 4.40 (8.27) | 11.50 (11.39)
  Percent change at Day 29 | 5.20 (9.94) | 7.80 (17.55)
  Percent change at Day 36 | 7.30 (7.64) | 8.80 (11.09)
  Percent change at Day 43 | 5.80 (7.73) | 11.60 (12.44)
  Percent change at Day 50 | 4.50 (5.77) | 3.50 (16.45)
  Percent change at Day 57: number analyzed (Participants) | 12 | 11
  Percent change at Day 57 | 3.40 (8.71) | 18.80 (7.84)
  Percent change at Day 64 | 0.80 (7.48) | 16.90 (14.18)

28. Secondary Outcome: Duration of Low Density Lipoprotein (LDL) Lowering Effects
Description: In this outcome measure duration of the lipid-lowering effects was reported. Lipid lowering was defined as decrease in LDL-C levels by greater than or equal to 15 percent.
Time Frame: Day 4 to Day 64
Population: Pharmacodynamic analysis population included all enrolled participants who received any amount of study medication and had at least 1 pharmacodynamic parameter of interest.
Measure: Median (Full Range); unit: days
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
days | 48.5 (16.36) [2.0 to 64.0] | 18.0 (15.68) [0.0 to 59.0]

29. Secondary Outcome: Number of Participants With Toxicity or Intolerable Dose Criteria
Description: Toxicity criteria included any of the following: serious adverse event; increased liver transaminases (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]: increased to greater than [>] 5*upper limit of normal reference range [ULN]); increased bilirubin (in absence of ALT or AST elevations, common terminology criteria for adverse events [CTCAE] greater than or equal to [>=] Grade 2); pancreatitis, increased serum creatinine (CTCAE >= Grade 2); creatine kinase, hyperglycemia or hypoglycemia, diarrhea or enteritis or nausea (CTCAE >= Grade 3); decreased platelet count (less than [<] 100000 per microliter); prolongation of QT interval with Fridericia's Correction (QTcF) (QTcF >500 millisecond [msec] [CTCAE >= Grade 3] or increase from baseline of >=60 msec) and other considered appropriate by investigator. CTCAE Grade 4.0: Grade 1= mild; Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening consequences and Grade 5= death related to adverse event.
Time Frame: Day 1 up to Day 64
Population: Safety analysis population included all participants who met the study enrollment criteria and had received any amount of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

30. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 64 days that were absent before treatment or that worsened relative to pretreatment state. Adverse events included both serious and non-serious adverse events.
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants
  AEs | 12 | 11
  SAEs | 1 | 0

31. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 64 days that were absent before treatment or that worsened relative to pretreatment state. AEs were assessed for severity by CTCAE Grade 4.0: Grade 1= mild; Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening consequences and Grade 5= death related to adverse event. Categories with at least 1 participant were reported
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants
  Grade 1 AEs | 5 | 8
  Grade 2 AEs | 4 | 3
  Grade 3 AEs | 2 | 0
  Unknown | 1 | 0

32. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants
  AEs | 6 | 0
  SAEs | 0 | 0

33. Secondary Outcome: Number of Participants With Systemic Treatment Emergent Adverse Events Identified by Physical Examination
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 64 days that were absent before treatment or that worsened relative to pretreatment state. Complete physical examination was conducted to assess skin, ears, throat, cardiac, respiratory, gastrointestinal, and musculoskeletal systems for systemic AEs.
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

34. Secondary Outcome: Number of Participants With Systemic Treatment Emergent Adverse Events Identified by Vital Signs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 64 days that were absent before treatment or that worsened relative to pretreatment state. Vital sign parameters body temperature, blood pressure and heart rate were assessed to identify systemic adverse events. AEs (all causalities), treatment related AEs and CTCAE severity grades for AEs were reported. CTCAE Grade 4.0: Grade 1= mild; Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening consequences and Grade 5= death related to adverse event. Categories with at least 1 participant were reported
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants
  AEs (All causalities) | 0 | 2
  Treatment related AEs | 0 | 0
  Grade 1 AEs: (All causalities) | 0 | 1
  Grade 2 AEs: (All causalities) | 0 | 1

35. Secondary Outcome: Number of Participants With Systemic Treatment Emergent Adverse Events Identified by Electrocardiogram (ECG) Parameters
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 64 days that were absent before treatment or that worsened relative to pretreatment state. ECG parameters RR interval, PR interval, QRS complex, QT interval, [Bazett's Correction], QTcF interval [Fridericia's Correction] were assessed to identify systemic AEs. AEs (all causalities), treatment related AEs and CTCAE severity grades for AEs were reported. CTCAE Grade 4.0: Grade 1= mild; Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening consequences and Grade 5= death related to adverse event. Categories with at least 1 participant were reported.
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants
  AEs (All causalities) | 0 | 1
  Treatment related AEs | 0 | 0
  Grade 1 AEs: (All causalities) | 0 | 1

36. Secondary Outcome: Number of Participants With Systemic Treatment Emergent Adverse Events Identified by Laboratory Parameters
Description: Laboratory parameters alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, gamma glutamyl transferase, lactate dehydrogenase, albumin, hemoglobin, protein, amylase, creatine kinase, lipase, basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets, white blood cells, bicarbonate, chloride, potassium, sodium, bilirubin, blood urea nitrogen, c-reactive protein , calcium, creatinine, direct bilirubin, glucose, magnesium, phosphate, uric acid, hematocrit, partial thromboplastin time , prothrombin time, red blood cells , urine pH, urine specific gravity were assessed to identify systemic AEs. AEs (all causalities), treatment related AEs and CTCAE severity grades for AEs were reported. Same participant may be reported in more than 1 CTCAE severity grade. Categories with at least 1 participant were reported.
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants
  AEs (All causalities) | 2 | 1
  Treatment related AEs | 2 | 0
  Grade 1 AEs: (All causalities) | 0 | 1
  Grade 1 AEs: (Treatment related) | 2 | 0
  Grade 2 AEs: (Treatment related) | 1 | 0
  Grade 3 AEs: (Treatment related) | 1 | 0

37. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA)
Description: Human serum ADA samples of participants who received PF-04950615 (RN316) were analyzed for the presence of anti-PF-04950615 (RN316) antibodies. Results with titer value >=4.32 nanogram per milliliter of anti-PF-04950615 antibodies were counted as positive. Number of participants with presence of anti-PF-04950615 antibodies were reported in this outcome measure.
Time Frame: Day 1 up to Day 64
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Number analyzed (Participants) | 12 | 12
Participants | 4 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04950615 (RN316) 4 mg/kg + Atorvastatin | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04950615 (RN316) 4 mg/kg + Atorvastatin (N=12) | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin (N=12)
Headache (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04950615 (RN316) 4 mg/kg + Atorvastatin (N=12) | PF-04950615 (RN316) 0.5 mg/kg + Atorvastatin (N=12)
Palpitations (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Injection site erythema (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2
Hordeolum (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood amylase increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Heart rate increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 4 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
All determinations of primary or secondary outcomes were arbitrary as study did not specify primary or secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.